CLINICAL TRIAL: NCT06363994
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Phase 3 Study of Orelabrutinib in Combination with Rituximab and Bendamustine (BR) Vs. BR in Subjects with Treatment-Naїve Mantle Cell Lymphoma
Brief Title: A Global Phase 3 Study of Orelabrutinib+BR Vs.BR in Pts with TN MCL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InnoCare Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00128
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: Orelabrutinib; Drug: Bendamustine Injection; Drug: Rituximab
- Arm B (Active Comparator)
  Interventions: Drug: Bendamustine Injection; Drug: Rituximab; Drug: Orelabrutinib Placebo

INTERVENTIONS:
Drug: Orelabrutinib — Eligible patients will receive Orelabrutinib orally as per the protocol，until disease progression or other reasons for treatment discontinuation，whichever comes first.
  Arms: Arm A
Drug: Bendamustine Injection — Eligible patients will receive Bendamustine by injection as per the protocol
Drug: Rituximab — Eligible patients will receive Rituximab by injection as per the protocol
Drug: Orelabrutinib Placebo — Eligible patients will receive Orelabrutinib Placebo orally as per the protocol
  Arms: Arm B

SUMMARY:
Compare the efficacy and safety of Orelabrutinib plus bendamustine+ rituximab versus bendamustine + rituximab in previously untreated patients with mantle cell lymphoma (MCL)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 65 of age, or ≥ 60 and < 65 years old who are ineligible for stem cell transplant or have refused stem cell transplantation due to reason(s) including: Have not received prior systemic therapies for MCL.
2. Modified Ann Arbor stage II-IV. Patients with stage II require systemic treatment to be eligible, at the discretion of the investigator.
3. Histopathological confirmed MCL, expression of Cyclin D1 and/or t (11; 14) chromosomal translocation. Either fresh tissue or FFPE for diagnosis must be sent to central lab for final confirmation after randomization.
4. At least one measurable site of disease (the longest axis of the lymph node lesion is > 1.5 cm, or the longest diameter of the extranodal lesion is > 1.0 cm).
5. ECOG PS score of 0 to 2.

Exclusion Criteria:

1. Existing or prior history of other malignant tumor and no evidence of recurrence and metastasis within 2 years before screening.
2. Subjects with evident gastrointestinal dysfunction that may affect drug intake, transport or absorption, or subjects who have undergone total gastrectomy.
3. Subjects for whom the goal of therapy is tumor debulking prior to stem cell transplant.
4. Use of strong inhibitors or strong inducers of cytochrome P450 3A within 14 days or 5 half-lives, whichever is longer, before the first dose of study treatment; or plan to use strong inhibitors or strong inducers of CYP3A during the study.
5. Known central nervous system lymphoma.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2031-06-25 (Estimated); Study Completion 2032-06-25 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
Progression-free Survival (PFS) for Arm A vs. Arm B | Approximately 7 years

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - The First People's Hospital of Changzhou, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chongqinq Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The second Hospital of Dalian Medical University, Dalian
  - Fujing Cancer Hospital, Fuzhou
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang University Medical School affiliated to the first Hospital, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Shandong Provincial Hospital, Jinan
  - The First Affiliated Hospital of Ningbo University, Jinan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University, Nanjing
  - Cancer Hospital Affiliated to Fudan University, Shanghai
  - Huashan Hospital of Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - The Tumor Hospital Affiliated to Xinjiang Medical University, Ürümqi
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and, Wuhan
  - The First Affiliated Hospital of the PLA Air Force Military Medical University (Xijing Hospital), Xi'an
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi'an
  - Yibin Second People's Hospital, Yibin
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No